CLINICAL TRIAL: NCT06677268
Title: Benefit of Respiratory Rehabilitation on Objective Sleep Quality in Patients with Stable COPD
Brief Title: Respiratory Rehabilitation and Sleep Quality in COPD Patients
Acronym: REARSOM/BPCO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022/0347/HP
Record Dates: First submitted 2024-10-15; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: polysomnography; sleep quality; physical activity; education; respiratory rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Initiation and Maintenance Disorders; Motor Activity | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: randomized, controled, interventional, multi center
Who Masked: Investigator
Masking Description: Investigators analyzing the polysomnography and total sleep time (primary endpoint) will be blinded of the group in which the patient is randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- interventional (Experimental): Patient in this arm will perform a 2-months respiratory rehabilitation program
  Interventions: Procedure: rehabilitation
- control (No Intervention): patient in the control group will have standard care without respiratory rehabilitation program

INTERVENTIONS:
Procedure: rehabilitation — Patients will undergo a respiratory rehabilitation program (24 exercise sessions of 90 minutes each, three times a week for 8 weeks and up to 9 therapeutic education workshops of 1 hour of the patient's choice)
  Arms: interventional

SUMMARY:
COPD affects 5 to 8% of the population in France. The disease consists of inflammation of the large and small airways causing permanent obstruction of the airways and symptoms such as dyspnea, cough and sputum that worsens over time.

Among all COPD patients, 40% complain of sleep disorders. Polysomnography data showed a prolongation of sleep onset latency and a decrease in deep sleep, correlated with the severity of daytime hypoxemia. Conversely, poor sleep quality leads to an increase in dyspnea, altered quality of life and increased occurrence of COPD exacerbations.

Respiratory rehabilitation has demonstrated significant benefits on exercise capacity, dyspnea, COPD exacerbations and quality of life. To the investigators' knowledge, a few studies have investigated the relationship between physical activity and sleep quality using polysomnography in this population. Thus, the aim of the study is to evaluate the benefits of respiratory rehabilitation on sleep architecture in patients with COPD. Investigators' hypothesis is that a respiratory rehabilitation program would improve the quality of sleep measured by polysomnography. Therefore, patient with COPD and no exacerbation in the previous year will be randomly assigned to the interventional group who perform the rehabilitation program or to the control group who will not perform the program. The primary endpoint is the sleep quality estimated by total sleep time as measured by the mean of 2 independent polysomnography readings, at baseline and after the RR program in the interventional group and after 2 months of usual care in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ age 50
* COPD defined according to the GOLD 2022 criteria, clinically stable (without exacerbation for at least 4 weeks), with indication for respiratory rehabilitation
* Absence of respiratory rehabilitation in the past 12 months
* Patient affiliated to the social security system
* For women of childbearing potential who have been on effective contraception (estrogen-progestogen or intrauterine device or tubal ligation) for 1 month.
* For postmenopausal women: confirmatory diagnosis (non-medically induced amenorrhea for at least 12 months prior to the inclusion visit)
* Patient who has read and understood the information letter and signed the consent form

Exclusion Criteria:

* BMI≥ 30 kg/m2
* Previously documented OSA (AHI > 10/h)
* Patient with a CPAP or NIV
* Patient on systemic corticosteroid therapy
* Patient on centrally acting therapy (benzodiazepine or opiate)
* Patient with an occurrence of severe COPD exacerbation
* Patient with other associated chronic respiratory insufficiency
* Patient with active cancer
* Patient with neuromuscular disease
* Patient with an osteoarticular disability or traumatic or neurological sequelae preventing participation in the respiratory rehabilitation program
* Psychiatric, cognitive or linguistic disorders with inability to understand to follow the protocol
* Patient with a contraindication to respiratory rehabilitation or any pathology preventing physical rehabilitation
* Patient with a cardiovascular contraindication to respiratory rehabilitation
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial safeguard, guardianship or curatorship
* Person subject to a legal protection measure
* Pregnant or parturient or breastfeeding woman

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Total sleep time (TST) | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  measured by the average of the 2 independent polysomnography scorings

SECONDARY OUTCOMES:
Sleep onset latency | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  Sleep onset latency (SOL) measured by the average of the 2 independent polysomnography readings
Pittsburgh sleep quality index (PSQI) | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  subjective sleep quality measured by the questionnaire PSQI
Quality of Life | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  measured by Saint George's Hospital Respiratory Questionnaire (SGRQ)
Daytime sleepiness | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  measured by Epworth Sleepiness Scale
Dyspnée | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  measured by the score modified Medical Research Council [mMRC]
Severity of COPD symptoms | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  measured by COPD Assessment Test [CAT]
Anxiety and depression | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  measured by the HAD (Hospital Anxiety and Depression) scale
exercise capacity | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  measured during an maximal exercise test
6 minutes walking test | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group
  measured by distance walked during 6 minutes.
Wakefulness after sleep onset | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  Wakefulness after sleep onset (WASO) measured by the average of the 2 independent polysomnography readings
Sleep Efficiency | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  Sleep Efficiency measured by the average of the 2 independent polysomnography readings
Number of awakenings | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  Number of awakenings measured by the average of the 2 independent polysomnography readings
Micro-arousal index | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  Micro-arousal index measured by the average of the 2 independent polysomnography readings
N1 sleep stage | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  N1 (%) measured by the average of the 2 independent polysomnography readings
N2 sleep stage | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  N2 (%) measured by the average of the 2 independent polysomnography readings
N3 sleep stage | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  N3 (%) measured by the average of the 2 independent polysomnography readings
other sleep parameter | at baseline and after the respiratory rehabilitation program in the interventional group (2.5 months) and after 2 months of usual care in the control group.
  REM (%) (Rapid Eye Movement) measured by the average of the 2 independent polysomnography readings

IPD SHARING:
Plan to Share IPD: Undecided